CLINICAL TRIAL: NCT00478296
Title: Case Report: Resolution of Pulmonary Hypertension With Sildenafil and Bosentan in Patients With Trisomy 21 and Atrial Septal Defect
Brief Title: Pulmonary Hypertension in Trisomy 21 Patients
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Other Study IDs: 07-021
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2008-01

CONDITIONS: Congenital Disorders
Keywords: Pulmonary hypertension; Sildenafil; Bosentan; Trisomy 21; Atrial septal defect
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Hypertension, Pulmonary; Down Syndrome; Heart Septal Defects, Atrial

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evidence has shown poor outcome for adult patients with pre-operative pulmonary hypertension following closure of an atrial septal defect. Life-threatening pulmonary hypertensive crises may occur in these patients when they no longer have an atrial communication to decompress high right heart pressures. This concern has led some to advocate fenestrated patch closure of ASDs in patients with pulmonary hypertension with the prospect of a repeated procedure in order to close the fenestrations at a later date.

DETAILED DESCRIPTION:
Pre-operative resolution of pulmonary hypertension would clearly provide the best long-term outcome for these patients, allowing a definitive surgical procedure. There are no reported cases of resolution of pulmonary hypertension with the use of pulmonary vasodilators allowing successful ASD closure.

We report the case of a patient with trisomy 21 and a primum atrial septum defect with associated cleft mitral valve who was diagnosed with pulmonary hypertension at 8 days of life. Elevated pulmonary pressures were documented by cardiac catheterization during which the patient was found to have minimally responsive pulmonary vasculature to the administration of oxygen. He was started on pulmonary vasodilators which were continued for the following 5 months which resulted in gradual reduction in estimated PA pressure allowing successful closure of the primum ASD and repair of the cleft mitral valve. Following surgery, he was not restarted on pulmonary vasodilators and has continued to do well. The ability to reverse his pulmonary hypertension through the use of pulmonary vasodilators made him a candidate for his successful, definitive surgical repair. He currently has no residual cardiac problems and requires no cardiac medications. There will be no patient follow-up.

ELIGIBILITY:
Inclusion Criteria:

* case report of a patient with trisomy 21 and primum atrial septum defect with associated cleft mitral valve who was diagnosed with pulmonary hypertension at 8 days of life

Exclusion Criteria:

* those who do not fit into inclusion criteria

Max Age: 8 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a case report of one subject with trisomy 21 and a primum atrial septum defect with associated cleft mitral valve who was diagnosed with pulmonary hypertension at 8 days of life.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2004-10; Primary Completion 2007-02 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Phelps, DO, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States